CLINICAL TRIAL: NCT01420523
Title: Phase II Pilot Study Evaluating the Efficacy of Dual Therapy With Raltegravir Plus Maraviroc in Patients Receiving Suppressive Antiretroviral Therapy and Presenting With Lipohypertrophy (ANRS 157 ROCnRAL).
Brief Title: Evaluation of Raltegravir Plus Maraviroc Therapy in Controlled HIV Patients Presenting With Lipohypertrophy
Acronym: ROCnRAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-002483-24
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Human Immunodeficiency Virus; Lipohypertrophy
Keywords: HIV; Lipohypertrophy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir-Maraviroc (Experimental): Raltegravir 400 mg twice a day + Maraviroc 300 mg twice a day
  Interventions: Drug: Raltegravir-Maraviroc

INTERVENTIONS:
Drug: Raltegravir-Maraviroc — Raltegravir 400 mg twice a day + Maraviroc 300 mg twice a day
  Other Names: Isentress and Celsentri

SUMMARY:
Evaluation of antiretroviral therapy combining Raltegravir and Maraviroc in patients with virological success, presenting with clinical lipohypertrophy.

DETAILED DESCRIPTION:
Assess the ability to maintain the plasma HIV viral load below the threshold needed for detection (< 50 copies/mL) at 24 weeks of raltegravir/maraviroc therapy without NRTIs and PIs, in patients with virological success and presenting with clinical lipohypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV-1 type B or CRF02.
* ≥ 18 years old
* Patients who have been receiving antiretroviral therapy for at least 5 years, and whose treatment has been stable for at least 6 months.
* Patients whose plasma viral load has been undetectable (below 200 copies/mL) over the last 24 months, and < 50 copies/mL for at least 12 months.
* Patients with an R5* tropic virus, as determined through DNA and with CD4 nadir ≥ 100/mm3
* Patients presenting with clinical lipohypertrophy recognized by themselves and by their doctors, and defined by increased volume of the abdominal and/or thoracic and/or cervical area (buffalo hump).
* Patients who have never been treated with raltegravir.
* Patients who have never been treated with maraviroc.
* Efficient contraception for women
* Free and informed written consent, signed by the patient and the investigator.
* Patients with health insurance. * To increase the certainty of selecting patients with an R5 virus, the HIV-1 tropism will be determined by the genotype method and interpreted with the Geno2pheno[coreceptor] algorithm and a false positive rate threshold for X4 virus at 20%, rather than the usual 10%.

Exclusion Criteria:

* X4, X4/5 or undetermined tropism of the HIV virus.
* HIV-2 or coinfection HIV-1/HIV-2.
* Chronic viral hepatitis B.
* Chronic viral hepatitis C requiring specific treatment over the first 24 weeks.
* Treatment with growth hormones.
* Hypolipemic or diabetes treatment, begun within the last 3 months.
* Pregnant or breastfeeding women.
* Haemoglobin < 7g/dl, neutrophils < 500/mm3, platelets < 50 000/mm3, creatinine clearance < 50 mL/min, alkaline phosphatases, ASAT, ALAT or bilirubin ≥ 3 times the upper limit of the normal range (N).
* Antiretroviral treatment associated to enzymatic inducer.
* Chronic alcohol consumption.
* Subjects under "sauvegarde de justice" (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship.
* Subjects participating in another clinical trial evaluating different therapies and including an exclusion period that is still in force during the screening phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Virological failure | Week 24
  Occurrence of virological failure, as verified by 2 consecutive plasma viral load measurements > 50 copies/mL, taken 2 to 4 weeks apart at most, during the first 24 weeks.

SECONDARY OUTCOMES:
Viro-immunological efficacy | Between baseline and W48
  * Proportion of patients with a HIV RNA viral load < 50 copies/mL.
  * Proportion of patients discontinuing the therapy:
  * Plasma genotypic resistance profile where the viral load is > 50 copies/mL.
  * Evaluation of DNA/RNA tropism in the event of failure.
  * Evaluation of plasma HIV RNA where the viral load is < 50 copies/mL, through ultrasensitive PCR testing.
  * Evolution of the CD4 and CD8 T-cell counts.
  * Blood concentration of raltegravir and maraviroc.
Tolerability criteria and metabolic impact | Between baseline and W48
  * Changes in glucose and lipid balance.
  * Changes in anthropometric measurements.
  * Number and severity of clinical and biological adverse effects.
  * Changes in bone mineral density and body composition, as measured by DEXA scan.
  * Changes in inflammation and endothelial activation markers between baseline and W48
  * Measurement of fat cells differentiation markers in adipose tissue biopsy samples
Compliance | Between baseline and W48
  • Assessment of compliance conducted at screening and at W24 and 48.
Quality of life | Between baseline and W48
  • Assessment of health-related quality of life conducted at baseline and at W24 and 48.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — Groupe hospitalier Pitié-Salpétrière; Dominique Costagliola, Study Director — Inserm U943
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

REFERENCES:
- [Derived] Soulie C, Assoumou L, Darty M, Rodriguez C, Donati F, Sayon S, Peytavin G, Valantin MA, Caby F, Schneider L, Canestri A, Costagliola D, Katlama C, Calvez V, Marcelin AG; ROCnRAL ANRS-157 Study Group. Virological factors associated with outcome of dual maraviroc/raltegravir therapy (ANRS-157 trial). J Antimicrob Chemother. 2015 Dec;70(12):3339-44. doi: 10.1093/jac/dkv280. Epub 2015 Sep 22. PMID 26396157
- [Derived] Katlama C, Assoumou L, Valantin MA, Soulie C, Duvivier C, Chablais L, Kolta S, Pialoux G, Mercie P, Simon A, Costagliola D, Peytavin G, Marcelin AG; ROCnRAL ANRS 157 Study Group. Maraviroc plus raltegravir failed to maintain virological suppression in HIV-infected patients with lipohypertrophy: results from the ROCnRAL ANRS 157 study. J Antimicrob Chemother. 2014 Jun;69(6):1648-52. doi: 10.1093/jac/dkt536. Epub 2014 Feb 16. PMID 24535278
- See also: Related Info — http://www.anrs.fr